CLINICAL TRIAL: NCT06150508
Title: Randomized Controlled Trial of the Smart Online-to-Offline Model Development for Chronic Diseases Management Through Digital Health in Real World Setting
Brief Title: Randomized Controlled Trial of the Smart O2O Model Development for Chronic Diseases Management Through Digital Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korea Health Industry Development Institute (Other Government); Seoul National University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB No: 2308-183-1463
Record Dates: First submitted 2023-11-09; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Hypertension; Diabete Mellitus
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparative group (No Intervention): Comparators will not be provided with the O2O service, but will be treated as usual (TAU) through the 1st tier health care clinics/centers in Pyeongchang-gun county.
- Intervention group (Experimental): Intervention group will use the service app "Value Health" for life-log recording. They regularly record life-log data such as blood pressure, blood glucose, medication, diet, exercise, and weight. (As mentioned, glucose level and blood pressure measurements will be automatically shared with the app using Bluetooth function of the provided checkers.) Interventions through application include automated message and alarm service through the app, as well as personalized intervention messages, record management, and other interventions from the Smart Healthcare Center and the primary healthcare provider.
  Interventions: Behavioral: O2O digital healthcare service

INTERVENTIONS:
Behavioral: O2O digital healthcare service — The O2O service includes a mobile app and web-based portal that allows patients to monitor their blood glucose levels, track their medication use and physical activity, receive personalized feedback and education, and communicate with healthcare providers. The treatment group will receive a blood sugar checker and blood pressure checker that send the records automatically to the application through Bluetooth.
  Other Names: O2O digital healthcare service for patients with diabetes and hypertension
  Arms: Intervention group

SUMMARY:
Objectives The aim of this intervention is to assess how well and how efficiently the O2O Service Model works in delivering primary healthcare and managing chronic diseases for patients living in Pyeongchang-gun at the local government level.

Trial design This is a randomized controlled trial with restricted, batch, blocked and individual random assignment. Investigators will allocate 1,000 participants from Pyeongchang-gun into two groups: one with diabetes (and pre-diabetes) and one with hypertension (including borderline cases), focusing on poorly controlled patients. As participants visit local health centers, their data will be sent to the research team for blocked randomization based on disease type, severity, and region. Assignment results will be communicated back to the centers and patients.

Study setting The intervention will take place in Pyeongchang-gun, Kangwon-do, South Korea. The Smart Healthcare Center affiliated to Public Medical Center of Pyeongchang will primarily manage the O2O service by providing necessary education and human resources while receiving and monitoring data from each participant and local medical centers. The overall study (including the design of trial) is managed by Seoul National University College of Medicine while the provision of O2O service and data collection are primarily in charge of Smart Healthcare Center of Pyeongchang.

Intervention in O2O Service Model:

After initial health exams, each patient gets a custom care plan, classifying their disease and care level. The Pyeongchang Smart Healthcare Center, with doctors, tracks patients via an online platform, sending automated health messages. High-risk patients receive a two-week glucose monitor and guidance on lifestyle adjustments. Doctors access patient health records through the participant's personal online datastore (POD), with consent, integrating health and prescription history from national insurance, and can assess heart disease risk.

Sample size The trial's sample size is determined using the MDES(Minimum Detectable Effect Size), with 1,000 participants divided equally between diabetes and hypertension groups. Each group is then split into treatment and control subgroups through random allocation. The MDES calculation, accounting for an explained outcome variation of 50% due to blocking and controls, and based on 500 subjects per group with equal allocation, aims for a high-accuracy effect size of 0.216 at a 5% significance level and 80% power.

Assignment of interventions: allocation Participants will be randomly placed into groups by a computer program. This study uses a specific randomization method that is restricted and organized by individual characteristics. The research team will tell the centers and patients about their group assignment via phone and email. Neither the healthcare staff nor the participants will know the group allocation beforehand. The research team is in charge of the randomization process and informing everyone involved. The staff at Pyeongchang's Smart Healthcare Center will sign up participants and manage their placement into the assigned intervention groups. There will be no blinding after participants are assigned to their groups.

List of Data For the study, the investigators have created questionnaires and interview formats to collect various data types, including random assignment records, baseline information, outcomes, service usage and costs, demographic and health details, physician-collected health records, life-log data from apps or web, clinical exam results, and service effectiveness and efficiency from the perspective of medical staff and administrators.

Statistical methods For the analysis of primary and secondary outcomes, the investigators will employ ITT(Intention-to-Treat) and Regression-Adjusted Impact Estimate. When data allows (especially data from control group), the investigators will also conduct timeseries effect analysis. To investigate the time-series changes in program effects across multiple time points, the dependent variable (outcome variable) should be measured at each time point to estimate program effects repeatedly.

Data management and monitoring The data management for the study will be conducted using electronic systems for secure and accurate data entry, coding, and storage, with robust checks and backups to ensure data quality, which will be archived for three years in compliance with bioethics standards before disposal according to privacy regulations. Participant confidentiality is prioritized through secure data collection and restricted access, with sharing only to authorized research team members and regulators using password protection or encryption. Additionally, a dedicated Data Monitoring Committee will oversee trial progress and adherence to protocols, while the Smart Healthcare Center collaborates with healthcare workers to manage patient services, with minimal adverse events expected.

DETAILED DESCRIPTION:
Objectives The objective of this intervention is to evaluate the effectiveness and efficiency of the Online-to-Offline(O2O) Service Model developed to provide primary healthcare and management of chronic diseases targeting patients residing in Pyeongchang-gun at the local government level.

The randomized controlled trial of this intervention will help verifying the model, and provide valuable information about the effectiveness of an O2O digital healthcare service for patients with diabetes and hypertension. If the intervention is found to be effective, it has the potential to improve access to care and self-management for patients, which could lead to improved health outcomes and reduced healthcare costs. The implications from this study can also serve as credible evidence for decision making for provision of digital health care services in other regions of Korea as well.

Trial design This is a randomized controlled trial with restricted, batch, blocked and individual random assignment. For sampling before randomization, investigators plan to recruit two target disease groups in Pyeongchang-gun: one group with diabetes patients (including pre-diabetes patients), and another with hypertension patients (including borderline hypertension patients). Total 1,000 participants (500 per group) will be recruited, and the investigators plan to prioritize the poorly controlled patients when recruiting.

Primary mode of sampling is voluntary based, where patients sign up through the advertisement, promotional campaign, or information provided by the physicians. Some patients will be recommended and informed to join this trial by their physicians while promotional/advertising materials will be posted at participating medical centers((i.e., Pyeongchang Public Medical Center and local private clinic, local private medical centres in Pyeongchang) and the Pyeongchang official website. Flyers will also be distributed through voluntary village health supporting groups-named Village Health Committee. In the meantime, for patients who have already diagnosed to have diabetes and hypertension will also be recruited from participating medical centres in Pyeongchang (i.e., local medical centres, Pyeongchang Public Medical center).

When eligible patients who are willing to participate in this study visits local health centre for clinical tests, their data will be periodically sent to the research team to carry out blocked random assignment (block: disease, severity, region). The assignment results are notified to the centre/clinic and then to the patients. The allocation ratio is 1:1 for each disease (hypertension and diabetes).

Study setting The intervention will take place in Pyeongchang-gun, Kangwon-do, South Korea. (Pyeongchang-gun is a county in the province of Gangwon-do, South Korea. It is in the eastern part of the province with a population of around 43 thousand people estimated in 2020.) The Smart Healthcare Center affiliated to Public Medical Center of Pyeongchang will primarily manage the O2O service by providing necessary education and human resources while receiving and monitoring data from each participant and local medical centers.

As mentioned, the intervention targets patients (and borderline patients) in Pyeongchang, and the data is collected from participating patients through the device and application as well as from the local medical centers when patients participate in (both control and treatment group) regular follow-ups.

The overall study (including the design of trial) is managed by Seoul National University College of Medicine while the provision of O2O service and data collection are primarily in charge of Smart Healthcare Center of Pyeongchang. There are stakeholders to develop and manage the O2O model (specifically the mobile application, data platform), such as Kangbuk Samsung Hospital, Huray and DKI, and Seoul National University Hospital as well as XAIMED are in charge of managing the Public Health HRecord (PHR) data collected from the patients and local medical centers.

Interventions

Intervention in O2O Service Model:

Following baseline comprehensive health examinations, each participant's primary attending physician will develop an individualized care plan. This care plan includes identifying the representative disease group (diabetes, pre-diabetes, hypertension, borderline-hypertension) and determining the intensity of care (intensive or standard). In cases where participants have both diabetes and hypertension, they are categorized as diabetes patients. Participants with poorly controlled diseases (systolic blood pressure exceeding 140 or diastolic pressure over 90 in the hypertension group, and HbA1c levels exceeding 6.5% in the diabetes group) are assigned to the intensive care group. However, these classifications can be adjusted as necessary based on the patient's clinical condition.

The Pyeongchang Smart Healthcare Center, in collaboration with physicians, continuously monitors and intervenes as needed. Monitoring occurs through the administrator's web page of the O2O service platform, allowing oversight of the life-log data of the intervention group. Enrolled patients receive interventions in the form of automated or manual messages.

- Message Delivery through the Application: Personalized Educational Material: The content of these messages is determined based on the participant's baseline evaluation results. They consist of publicly available videos produced by reputable organizations, including academic societies, and are provided via links to YouTube videos.

Health Reports: Sent every three months, these reports provide a comprehensive evaluation of whether the individual's condition is being well managed based on life-log data from the past three months.

Manual Messages (Texted Messages): Indicator-based personalized messages are manually transcribed, evaluating the state of health management over the last two or four weeks based on life-log data. These messages are primarily drafted by the Pyeongchang Smart Healthcare Center, using pre-made message templates created by healthcare experts (doctors, nutritionists, nurses, etc.) suitable for each situation. Messages are sent to patients after final confirmation by their respective primary physicians. Additional messages can be sent as needed during the monitoring process, especially if blood pressure or blood glucose levels are at cautionary or dangerous levels or if data entry is insufficient.

- Continuous Glucose Monitor (Among the Intervention Group): Some diabetes patients in the intervention group will be provided with a continuous glucose monitor (Freestyle Libre). Eligibility for this monitor is determined based on their recorded glucose levels not reaching the normal range in more than half of their recent examinations within the latest 14 days. Patients eligible for the continuous glucose monitor receive notifications via text or phone call from the Smart Healthcare Center. They are required to attach the device for two weeks and are advised to self-monitor their glucose variations. During this period, they are strongly encouraged to manage their glucose levels by adapting their usual lifestyle. Some patients may receive the monitor again, if needed, two weeks after the detachment of the device.

- Personal Health Record (PHR) Data: PHR data can be accessed and utilized exclusively by attending physicians with patient consent through the participant's personal online datastore (POD) web view in the clinic. POD can import health screening results, medical history, and prescription history provided by the National Health Insurance Service (NHIS), which is mandatory for all citizens to enroll in. Additionally, POD contains AI-based retinal image analysis capable of detecting ophthalmologic abnormalities (e.g., glaucoma, diabetic retinopathy) and predicting cardiovascular disease (CVD) mortality risk. It also includes another CVD incidence prediction model developed using national health screening data. With access to this PHR data, attending physicians can provide comprehensive consultations to patients regarding their CVD risk.

- Control Group: The control group will receive treatment as usual, which is the typical care provided to individuals without the additional interventions described above.

Strategies to improve adherence to interventions Patients will be regularly reminded to use the mobile-app to check up their medical conditions with mobile alarms, notifications and in-person notification from the Smart Healthcare Center of Pyeongchang Medical Center

Relevant concomitant care permitted or prohibited during the trial Treat of as usual (TAU) is allowed for both control and treatment group. However, the investigators believe that patients' participation in alternative services will be the most difficult problem to solve during the study. The investigators have identified 'participating in another research program involving smart health technology' as one of the exclusion criteria. will not be eligible for inclusion in our study. At the same time, the investigators will further prevent concomitant care (that might be possible during the intervention) through information provision and by educating the operators who will be in charge of training and informing the patients for service utilization

Sample size Sample size is calculated using MDES (Minimum Detectable Effect Size) equation. The sample size for this study is determined with the aim of detecting a meaningful difference between the treatment and control groups with sufficient statistical power. Given that the total sample size is 1000 participants, the investigators will divide this cohort into two main groups: participants with diabetes and those with hypertension. Subsequently, each of these two groups will be randomly allocated into treatment and control subgroups. Calculation of MDES is separately carried out for the diabetes and hypertension groups, taking into account the unique characteristics and expected effect sizes within each group.

Assuming that the variation in the outcome variable that can be explained by blocked random assignment and control variable is about 50%, and assuming a sample of 500 subjects with a 5:5 allocation ratio, with a statistical significance level of 5% and a power of 80%, the MDES is 0.216. If the investigators assume that the variation in the outcome variable that can be explained by blocked random assignment and control variable is about 25%, the MDES is 0.187, which is still high in accuracy. Assuming that the variation in the outcome variable that can be explained by blocked random assignment and control variable is about 10%, the MDES is 0.181, which is still high in accuracy. (Note: Cohen (1988) suggested that an MDES of 0.20 is a small effect size, 0.50 is a medium effect size, and 0.80 is a large effect size.) Therefore, the investigators aim to recruit the sample of 500 participants for each disease type, and the treatment-to-control ration is 5:5 for each disease group

Recruitment There are two concurrent recruitment procedures, each with slight distinction. Procedure 1 primarily targets patients previously diagnosed with diabetes, pre-diabetes, hypertension, or borderline hypertension. Procedure 2 targets respondents who have been exposed to our promotion and advertisement efforts. For these respondents who voluntarily asked to enroll, their eligibility will be confirmed when they are either: 1) Previously diagnosed with diabetes, borderline diabetes, hypertension, or borderline hypertension (with proof of diagnosis) or 2) Newly diagnosed with any of these conditions through the comprehensive health check-up included in this intervention procedure.

Assignment of interventions: allocation Sequence generation Participants will be randomized using a computer-generated randomization sequence. This study will apply a restricted, batch, blocked, individual random assignment. After screening the participant eligibility, each eligible participant will be contacted to receive informed consent. For those who consented to participate will visit the local medical center (or smart healthcare center) for detailed explanation of service, to physically signed the agreement, receive training to use the mobile app, and respond the survey. After patients receive clinical tests at the clinic, the list of patients and test results are periodically sent to the research team. The research team conducts blocked random assignment periodically based on disease, severity, and region. The assignment results are notified to the center and clinic and then to the patients by the research team. Such process is designed to align to the O2O service process.

Concealment mechanism Mechanism of implementing the allocation sequence is using central telephone and email. The health care staffs and participants won't know the allocation until the research team inform them.

Implementation The research team will generate the allocation sequence, deliver the allocation results to the center and patients directly. The staffs of Smart Healthcare Center of Pyeongchang Public Medical Center will enroll participants and assign participants to interventions.

Assignment of interventions: Blinding Who will be blinded Once the random assignment is conducted, no blinding will take place for this study.

Data collection and management Plans for assessment and collection of outcomes

Data Quality Assurance:

To ensure the integrity of our survey data, the investigators have implemented several processes to promote data quality. First, the investigators plan to employ duplication risk mitigation measures by cross-referencing participant phone numbers and birth dates. This step helps identify and rectify any duplicate entries, maintaining the accuracy and uniqueness of our dataset.

Second, our assessors will be rigorously trained to conduct surveys effectively. The investigators have developed a comprehensive manual guide to standardize data collection procedures. This guide serves as a valuable resource for our assessors, ensuring consistency and adherence to established protocols.

Furthermore, prior to the commencement of the intervention, the assessors will also undergo a pre-intervention session. During this session, they will receive training on data collection processes, ensuring their familiarity with survey instruments and questionnaires.

Additionally, our Smart Healthcare Center plays a pivotal role as a call center, promptly addressing any issues or queries that may arise during data collection. This continuous support mechanism helps maintain data quality throughout the study.

Study Instruments:

For data collection, the investigators have developed survey questionnaires and interview guides. These instruments have been meticulously crafted, drawing from health outcome indicators aligned with clinical guidelines. This alignment ensures that our data collection tools are both relevant and comprehensive, enabling us to capture essential information related to our study objectives.

Our commitment to data quality and the robustness of our study instruments underpins the reliability and validity of the data collected, ensuring the credibility of our research findings.

List of Data Data to be collected for this study can be categorized into 'Record of Random 'Assignment,' 'Baseline,' 'Outcome,' 'Service Utilization data,' 'Service Cost Data'.

Plans to promote participant retention and complete follow-up

The research team's strategy to retain the completeness of random assignment while managing any contamination or drop-out is the following:

* Conduct a pilot random assignment for about a week to identify any issues.
* Continuously check the size of Treatment group (T) and Comparison group © considering the sample size by group to monitor the possibility of non-random assignment.
* Issue of random assignment of ineligible applicants: If found in both T and C, they will be dropped from the sample; if found only in T, no-show adjustment will be made at the analysis stage.
* Control group contamination:

  1. Identify Contamination by participants vs. contamination by operators
  2. Education for operators
  3. Minimizing face-to-face contact between operators and participants
  4. Direct notification of random assignment results to participants by the research team
* Cross-over: When the controller applies for random allocation again. Do not remove from the sample, but handle as no-show adjustment at the analysis stage.

The field operators (i.e., staffs of Smart Healthcare Center and Public Medical Center of Pyeongchang) will regularly check-up with the patients to remind them to use the mobile application, while the patients will be automatically notified via app notification and e-mails for service use. When participants request discontinuation, they will be asked to fill out the follow-up survey and their medical records (from medical centers and National Health Insurance Service) will be collected at the point of discontinuation. For deviated participants, medical records (from medical centers and National Insurance Service) will be collected when the deviation is identified.

Data management

The data management plan is the following for each process:

Data entry: All data will be entered using electronic data capture (EDC) software. Two independent operators will perform double data entry for accuracy.

Coding: A coding manual will be created to ensure consistency in coding. All coded data will be verified by a second operator for accuracy.

Security: Access to the data will be password-protected, and only authorized personnel will have access. The data will be stored on a secure server that is regularly backed up.

Storage: The data will be stored in an electronic format. The data will be stored on a secure server located within the research institution.

Data quality processes: Range checks will be performed to ensure that data values fall within acceptable ranges. Data cleaning procedures will be performed to correct any discrepancies or missing data. The final dataset will be verified for completeness and accuracy by the research team before analysis.

Backup and archiving: The data will be regularly backed up to ensure its integrity in case of system failure or loss. A copy of the final dataset will be archived in a secure location for future reference. According to Article 15 of the Enforcement Rules of the Bioethics and Safety Act, all research-related records and data will be archived for three years from the end of the research.

Data Disposal: Seoul National University, an institution that is in charge of retention, will dispose of any data and document containing personal information in accordance with Article 16 of Enforcement Decree of the Personal Information Protection Act after three years of archiving.

Confidentiality

The investigators will collect personal information about potential and enrolled participants through informed consent forms, medical records, and questionnaires. The investigators will ensure that all personal information is securely stored and accessed only by authorized personnel. The investigators will share personal information only with the research team and regulatory agencies, and the investigators will do so through password-protected access or encryption to ensure confidentiality.

The specific protocols are as follows:

The participant is provided with sufficient explanation and, if voluntarily agreed, signs a written consent form to participate in the research.

Confidentiality will be maintained for information that can identify the personal information.

Information can be provided if the participant inquires about the test results. The participant's data file will be stored on the server of the data management personnel. This server is accessible only to the principal investigator, research staff, and co-researchers, and the file is encrypted. Therefore, access is not possible except for those who participated in this research.

The data file collected during the research process will be provided to a third party (National Health Smart Management Research and Development Division under the Ministry of Health and Welfare, Government of South Korea) and submitted to the data platform (big data and personal data repository) established by the division. In this process, personal information is protected by applying the integrated authentication system and DID (Decentralized Identifier, a distributed identification technology based on blockchain technology) system developed by the division.

Statistical methods For the analysis of primary and secondary outcomes, the investigators will employ ITT(Intention-to-Treat) and Regression-Adjusted Impact Estimate.

When data allows (especially data from control group), the investigators will also conduct timeseries effect analysis. The occurrence of program effects and how these effects change over time are crucial pieces of information to be derived from this experimental study. Analysing the temporal trajectory of program effects is essential, as the timing of impact and the nature of the program can result in diverse patterns of change based on the severity of disease or behavioural patterns of patients.

In randomized experiments, comparability between randomly assigned program and control groups remains consistent over time. Therefore, analysing the time-series changes in program effects can be achieved by applying cross-sectional analysis methods (i.e., Equation (1)) at each time point. To investigate the time-series changes in program effects across multiple time points, the dependent variable (outcome variable) should be measured at each time point to estimate program effects repeatedly. It's important to note that, in Equation (1), the variables that change over time are the dependent variables only, while program variables and control variables remain constant. This is because, the distinction between program and control groups should not change over time, and control variables should be obtained prior to random allocation.

An important consideration for this analysis is that the "time" mentioned is relative, not absolute. It is measured relative to the random assignment date, not an absolute calendar year. Therefore, evaluators will record the random assignment date for all sample members and integrate it into the analysis dataset. The dependent variables obtained from administrative statistical databases should also be transformed into relative time variables based on the random assignment date for analysis.

Methods in analysis to handle protocol non-adherence and any statistical methods to handle missing data

Defiers in the Treatment Group: In the event that there is non-adherence to the protocol, particularly if there are individuals who defy the assigned treatment, the investigators will estimate the Local Average Treatment Effect (LATE). Since the control group will not be provided with the application, there is no possibility of 'defiers' in the control group. Therefore, the investigators will simply divide the ITT with the rate of compliers.

LATE= ITT/(Rate of Compliers (in Treatment Group)) To address missing data for variables of interest, the investigators will use a missing-dummy approach, specifically employing dummy variable adjustment. This method involves creating dummy variables to account for missing data and subsequently including these dummy variables in our analysis as covariates. This approach allows us to compensate for missing data and maintain the completeness of our analysis while minimizing the impact of missing observations on our results.

Oversight and monitoring Composition of the coordinating centre and trial steering committee Composition and Roles of Key Entities: The O2O service is orchestrated by a collaborative effort between the "Smart Healthcare Center" personnel and healthcare professionals situated at each patient's primary care clinic. The Smart Healthcare Center operates under the umbrella of the Public Health Center (PHC) of Pyeongchang-gun and comprises our dedicated team of researchers alongside PHC staff members.

Composition of the data monitoring committee, its role and reporting structure The Data Monitoring Committee (DMC) comprises members from the evaluation team, ensuring a diverse range of expertise to oversee the trial's data and processes. The Data Monitoring Committee plays a pivotal role in maintaining the integrity and quality of trial data. Its responsibilities include monthly monitoring and feedback sessions to assess the trial's progress and adherence to protocols. The Data Monitoring Committee reports its findings directly to the Principal Investigator (PI), providing valuable insights and recommendations to enhance the trial's efficacy and safety.

Importantly, the Data Monitoring Committee operates independently from the intervention itself. Its members do not have direct involvement with participating medical centers and the Pyeongchang Smart Healthcare Center. This independence ensures unbiased evaluation and decision-making regarding the trial's progress and safety.

Adverse event reporting and harms The likelihood of adverse events or unintended effects related to trial interventions or trial conduct is not anticipated to be high. However, in the event that such occurrences do arise, our response protocol is well-established. Any solicited or spontaneously reported adverse events will be promptly reported to the Principal Investigator (PI) overseeing the trial. Simultaneously, these events will be reported to the Seoul National University Hospital (SNUH) Institutional Review Board (IRB) Committee, the regulatory body responsible for overseeing the ethical and safety aspects of the trial. Upon notification of an adverse event or unintended effect, relevant and appropriate actions will be taken in response. These actions may include further investigation, adjustments to trial conduct, or any necessary modifications to ensure participant safety and the integrity of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Participation aged 18 to 70 years
2. Participation diagnosed with diabetes (including borderline diabetes) or hypertension (including borderline hypertension)

However, we will exercise flexibility in age eligibility, allowing patients above 70 years to participate if they meet the following criteria:

Digital Literacy: Participants above 70 years must demonstrate proficiency in digital technology and the ability to effectively use the mobile application "Value Health," which has been specially developed for this research.

Exclusion Criteria:

1. Incompatible Mobile Device: Individuals using older mobile phones that are not compatible with the "Value of Health" application will be excluded.
2. Participation in Concurrent Research: Individuals who are currently participating in another research program involving smart health technology will not be eligible for inclusion in our study.
3. Non-Acceptance of Random Assignment or Participation: Individuals who do not agree to be randomly assigned to either the treatment or control group or who do not wish to engage in our research program will be excluded from participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Once each at baseline for all participants, and 6 months after for hypertension patient or 9 months after for diabetes patient (Total 2 times)
  Diastolic blood pressure, Systolic blood pressure (mmHg)
Fasting blood glucose level (FBG) in mg/dL | Once each at baseline for all participants, and 6 months after for hypertension patient or 9 months after for diabetes patient (Total 2 times)
  Glucose level
Glucose level | Once each at baseline for all participants, and 6 months after for hypertension patient or 9 months after for diabetes patient (Total 2 times)
  HbA1c in percent
Lipid profile | Once each at baseline for all participants, and 6 months after for hypertension patient or 9 months after for diabetes patient (Total 2 times)
  Cholesterol, Triglyceride(TG), HDL Cholesterol, LDL Cholesterol(All in ㎎/㎗)

SECONDARY OUTCOMES:
Body measurement | Once each at baseline for all participants, and 6 months after for hypertension patient or 9 months after for diabetes patient (Total 2 times)
  Weight in kilogram, height in meters, BMI kg/m^2
Waist circumference in centimeter | Once each at baseline for all participants, and 6 months after for hypertension patient or 9 months after for diabetes patient (Total 2 times)
  Body measurement
Medication Adherence | Once each at baseline for all participants, and 6 months after for hypertension patient or 9 months after for diabetes patient (Total 2 times)
  Duration of Medication Use/Prescription Period
Costs of treatment (Healthcare expenditure) | up to 6 months after for hypertension patient or 9 months after for diabetes patient
  Healthcare expenditure related to manage the designated disease
Lifestyle questionnaire | Once each at baseline for all participants, and 6 months after for hypertension patient or 9 months after for diabetes patient (Total 2 times)
  We use questionnaire for assessing physical activity, smoking status and alcohol drinking. This questionnaire is based on Health checkup questionnaire for general health screening in Korea and Guideline for Primary Health Care Chronic Diseases Management Pilot Program(3rd Revision) in Korea. "In relation to physical activity, the assessment will include regular exercise habits, types of exercise, intensity of exercise, and the amount of exercise. Regarding alcohol consumption, current drinking status and drinking history will be evaluated. For smoking, lifelong smoking status, as well as current and past smoking history, will be confirmed.

OTHER OUTCOMES:
Participation rate | up to 6 months after for hypertension patient or 9 months after for diabetes patient
  Application utilization level (Daily or Weekly Active Users) in absolute user number and percent divided by all users, Record rate per user(percent calculated by all recorded day by all the study period)
Satisfaction rate | Once at 6 months after for hypertension patient or 9 months after for diabetes patient
  Satisfaction rate of doctors and care coordinators (by interview, in percent caculated by dividing satisfied doctors and care coordinators divided by all doctors and care coordinators), Patient satisfaction rate(by survey, in percent caculated by dividing satisfied of participants by all participants number)

CONTACTS AND LOCATIONS:
Overall Officials: Juwhan Oh, MD, PhD, Principal Investigator — Seoul National University Hospital & College of Medicine

IPD SHARING:
Plan to Share IPD: No
We will share personal information only with the research team and regulatory agencies, and we will do so through password-protected access or encryption to ensure confidentiality.

REFERENCES:
- [Derived] Shin JE, Choi J, Lee H, Lee SW, Oh J. Protocol paper: randomized controlled trial of the smart online-to-offline model development for chronic diseases management through digital health in real world setting. Trials. 2025 Feb 5;26(1):40. doi: 10.1186/s13063-025-08735-8. PMID 39910545